CLINICAL TRIAL: NCT07019272
Title: Efficacy and Safety of Neratinib as Extended Adjuvant Therapy in HER2-Positive Early Breast Cancer Patients Who Achieved pCR After Neoadjuvant Therapy But Have High-Risk Factors: A Multi-Center, Real-World Study From Hebei, China
Brief Title: Neratinib in Extended Adjuvant Treatment for HER2+ Early Breast Cancer With pCR But High-Risk Features: A Hebei Multi-Center Real-World Study
Status: Not yet recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025KY006
Record Dates: First submitted 2025-05-17; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Neratinib (HKI-272) — Sequential neratinib extended adjuvant therapy will be initiated within 6 months after completing standard trastuzumab-based adjuvant therapy, continuing for 1 year.
  As a real-world non-interventional study, treating physicians will determine neratinib regimens per the prescribing information and current clinical practice.
  Neratinib Dosing:
  Standard regimen: 240 mg (6 tablets) once daily with food for 1 year；
  Dose escalation (to mitigate diarrhea, per latest CSCO Breast Cancer Guidelines and FDA labeling):
  Week 1: 120 mg/day (days 1-7) Week 2: 160 mg/day (days 8-14) Week 3 onward: 240 mg/day (days 15-365)

SUMMARY:
Neratinib is an oral, irreversible pan-HER tyrosine kinase inhibitor. Current treatment guidelines recommend neratinib as an extended adjuvant therapy for HER2-positive breast cancer patients to further reduce the risk of recurrence.

Even when HER2-positive breast cancer patients achieve pathological complete response (pCR) after neoadjuvant therapy, those with high-risk factors (such as large tumors [cT3/T4] or lymph node-positive disease) still face a risk of cancer returning. However, there is limited data on the effectiveness and safety of neratinib in these patients.

This study aims to provide real-world evidence on how well neratinib works in high-risk HER2-positive breast cancer patients who achieved pCR, helping to improve treatment strategies for Chinese patients.

DETAILED DESCRIPTION:
This study is a single-arm prospective study with historical controls as external comparators

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, female
2. Clinical stage ≥cT3 or ≥cN1, regardless of hormone receptor (HR) status
3. HER2-positive: HER2 IHC 3+ or IHC 2+ with ISH+
4. Achieved pathological complete response (pCR) after neoadjuvant therapy
5. Completed 1 year of standard adjuvant therapy (including trastuzumab), with ≤6 months between the last adjuvant treatment and starting neratinib
6. No evidence of recurrence or metastatic disease (confirmed by clinical/imaging exams after completing standard adjuvant therapy and before starting neratinib)
7. Left ventricular ejection fraction (LVEF) ≥50%
8. ECOG performance status 0-1

Exclusion Criteria:

1. Hypersensitivity to any component of the investigational drug
2. Inability to swallow oral medication
3. Participation in another interventional clinical trial within 4 weeks before enrollment, or planned participation during this study
4. Use of any investigational drug within 14 days prior to treatment initiation
5. Concurrent chemotherapy, radiotherapy, immunotherapy, or biologic therapy for breast cancer
6. Severe psychiatric disorders preventing compliance with informed consent, treatment, or follow-up procedures
7. Pregnancy, lactation, or plans for pregnancy in the near future
8. Other significant medical conditions or laboratory abnormalities that, in the investigator's judgment, make participation unsuitable

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This study focuses on HER2-positive early breast cancer (EBC) patients who achieved pathological complete response (pCR) following neoadjuvant therapy but present with high-risk features (such as initial clinical stage cT3/T4 tumors or node-positive disease). These patients must have completed standard adjuvant therapy (including trastuzumab-based regimens) and initiated neratinib as extended adjuvant treatment within 6 months after completing their standard therapy.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease Free Survival (IDFS) | From Day 1 of treatment until 2 years after treatment completion
  IDFS, as defined by the STEEP System, was measured from the date of treatment to the date of first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence, regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, second primary non-breast invasive cancer, death attributable to any cause.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | From Day 1 of treatment until 2 years after treatment completion
  Disease-free survival is defined as the time from baseline until the first occurrence of DCIS or an iDFS event (an iDFS event including invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, or distant recurrence and death from any).
Overall Survival (OS) | From Day 1 of treatment until 2 years after treatment completion
  OS was defined as the time from baseline to death due to any cause, censored at the last date known alive.
Distant Disease-free Survival (DDFS) | From Day 1 of treatment until 2 years after treatment completion
  Distant disease-free survival time is defined as the time from baseline until the first occurrence of distant recurrence or death from any cause.
Time to distant recurrence | From Day 1 of treatment until the first distant tumor recurrence or metastasis
  defined as time from baseline to the date of the first distant recurrence or death from breast cancer
Cumulative incidence of CNS recurrence | From Day 1 of treatment until 2 years after treatment completion
Incidence of grade ≥3 diarrhea | From consent to 28 days after last dose
Incidence and severity of other adverse events (AEs) | From consent to 28 days after last dose
Treatment patterns of patients | From Day 1 of treatment until last dose

IPD SHARING:
Plan to Share IPD: No